CLINICAL TRIAL: NCT00197015
Title: Immunogenicity & Safety of GSK Biologicals' Inactivated Hepatitis A Vaccine (Havrix™) Co-administered With Merck & Company, Inc. Measles-Mumps-Rubella Vaccine (M-M-RII) & Merck & Co Varicella Vaccine (VARIVAX™) to Children 15 Months of Age
Brief Title: Immunogenicity & Safety of Hepatitis A Vaccine Co-admin With a Measles/Mumps/Rubella & a Varicella Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208109/231
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-04-01 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-10

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines; Chickenpox Vaccine

ARMS (3):
- HAV Group (Active Comparator): Subjects received 2 doses of Havrix® (1 dose at Day 0 and 1 dose between Month 6 and Month 9)
  Interventions: Biological: Havrix®
- HAV+MMR+V Group (Experimental): Subjects received 1 dose of Havrix®, coadministered with M-M-R®II and VARIVAX®, at Day 0 and 1 dose of Havrix® between Month 6 and Month 9
  Interventions: Biological: Havrix®; Biological: M-M-R®II; Biological: VARIVAX®
- MMR+V→HAV Group (Active Comparator): Subjects received 1 dose of M-M-R®II and VARIVAX® at Day 0 and then 2 doses of Havrix® (1 dose at Day 42 and 1 dose between Month 7.5 and Month 10.5)
  Interventions: Biological: Havrix®; Biological: M-M-R®II; Biological: VARIVAX®

INTERVENTIONS:
Biological: Havrix® — 2 doses administered intramuscularly
Biological: M-M-R®II — 1 dose administered subcutaneously
  Arms: HAV+MMR+V Group; MMR+V→HAV Group
Biological: VARIVAX® — 1 dose administered subcutaneously
  Arms: HAV+MMR+V Group; MMR+V→HAV Group

SUMMARY:
This is a study to evaluate the immune response and safety of GSK Biologicals 2-dose inactivated hepatitis A vaccine when administered with a measles/mumps/rubella vaccine and a varicella (chickenpox) vaccine in children as young as 15 months of age.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
An open, controlled comparison of Havrix™ administered alone or with MMR II and Varivax™. The three groups evaluated are: 1) Havrix™ alone, 2) Havrix™ + MMR II and Varivax™ and 3) MMR II and Varivax™ followed by Havrix™ one month later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents/guardians are believed by the investigator to be willing to comply with the requirements of the protocol
* A male or female child 12 and 13 months of age at the time of entry into the Enrollment Phase
* Written informed consent obtained from the parents or guardian of the subject,
* Free of obvious health problems as established by medical history and history-directed physical examination before entering into the study, and
* Parents/guardian of the subject must have a telephone or be able to be contacted by telephone

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 42 days preceding the first dose of study vaccine, or planned use during the study period, Chronic administration (defined as more than 14 days) of immuno-suppressant or other immune-modifying drugs within six months prior to vaccination or planned administration at any time during the study period. (For corticosteroids, this will mean prednisone, or equivalent, ≥0.5 mg/kg/day. Inhaled, nasal and topical steroids are allowed.) Planned administration or administration of any vaccine not foreseen by the study protocol during the period 31 days before and 31 days after each dose of study vaccine(s).
* Previous vaccination against hepatitis A,
* History of hepatitis A,
* Known exposure to hepatitis A,
* Previous vaccination against measles, mumps, rubella and/or varicella,
* History of measles, mumps, rubella and/or varicella,
* Known exposure to measles, mumps, rubella and/or varicella within 30 days prior to the start of the study,
* Planned chronic use of salicylates during the 6-week period following administration of the doses of study vaccine(s),
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection,
* A family history of congenital, hereditary or infectious immunodeficiency or parental risk factors for HIV infection,
* History of allergic disease/reactions or hypersensitivity likely to be exacerbated by any component of HavrixTM, M-M-RII or VARIVAXTM, including 2-phenoxyethanol, neomycin and gelatin,
* History of anaphylactic or anaphylactoid reactions to egg proteins,
* History of hypersensitivity/allergic reaction to latex. Note: The tip cap and the rubber plunger of the HavrixTM needleless pre-filled syringes contain dry natural latex rubber.
* Major congenital defects or serious chronic illness,
* Active untreated tuberculosis,
* History of significant blood dyscrasias
* History of any neurologic disorder (a history of febrile seizures not associated with an underlying neurological disorder does not exclude the subject)
* Acute disease at the time of vaccination
* Administration of immunoglobulins and/or any blood products within three months prior to the first dose of study vaccine or planned administration at any time during the entire study period

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1474 (Actual)
Dates: Start 2003-10-06; Primary Completion 2009-06-09 (Actual); Study Completion 2009-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (40):
  - GSK Investigational Site, Cabot, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Waukee, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Lumberton, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, University Heights, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Beaver Falls, Pennsylvania
  - GSK Investigational Site, Norristown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Rydal, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Rinderknecht S, Michaels MG, Blatter M, Gaglani M, Andrews W, Abughali N, Chandreshekaran V, Trofa AF. Immunogenicity and safety of an inactivated hepatitis A vaccine when coadministered with measles-mumps-rubella and varicella vaccines in children less than 2 years of age. Pediatr Infect Dis J. 2011 Oct;30(10):e179-85. doi: 10.1097/INF.0b013e31822256a5. PMID 21617573
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208109/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the total numbers of subjects enrolled in the study was 1474, the total number of subjects that entered the study was 1241. The remaining subjects received a subject number but no vaccine dose and were therefore excluded from the analysis and group assignment.
Period: Overall Study
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Started | 324 | 455 | 462
Completed | 274 | 366 | 385
Not Completed | 50 | 89 | 77
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 3
Not completed — Withdrawal by Subject | 17 | 37 | 34
Not completed — Lost to Follow-up | 28 | 46 | 37
Not completed — Other | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group | Total
Number analyzed (Participants) | 324 | 455 | 462 | 1241
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.0 (0.27) | 15.0 (0.22) | 15.0 (0.25) | 15.0 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 208 | 232 | 594
  Male | 170 | 247 | 230 | 647

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A Virus (HAV) Antibody Concentrations in HAV and HAV+MMR+V Groups.
Description: Concentrations are given as geometric mean concentrations (GMCs) expressed as milli-international units per milliliter (mIU/mL).
Time Frame: 31 days following the second dose of Havrix®
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results from HAV and HAV+MMR+V Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 206 | 0 | 286
mIU/mL | 1390.4 [1186.3 to 1629.6] |  | 1895.2 [1682.7 to 2134.5]

2. Primary Outcome: Number of Subjects With Anti-hepatitis A Virus (HAV) Antibody Concentration Equal or Above the Cut-off Value in HAV and HAV+MMR+V Groups
Description: Anti-HAV antibody cut-off value assessed include 15 milli-international units per milliliter (mIU/mL).
Time Frame: 31 days following the second dose of Havrix®
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 206 | 0 | 286
Participants | 204 |  | 285

3. Primary Outcome: Number of Subjects Seroconverted for Anti-measle, Anti-mumps and Anti-varicella Antibodies in HAV+MMR+V and MMR+V→HAV Groups
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination. Cut-off values assessed include 150 milli-international units per milliliter (mIU/mL) for anti-measles antibodies, 28 Effective Dose 50 (ED50) for anti-mumps antibodies and 1:5 for anti-varicella antibodies.
Time Frame: 42 days following the administration of M-M-R®II and VARIVAX®
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results from HAV+MMR+V and MMR+V→HAV groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 250 | 268
Participants
  Anti-measles |  | 247 | 267
  Anti-mumps: number analyzed (Participants) | 0 | 197 | 212
  Anti-mumps |  | 193 | 207
  Anti-varicella: number analyzed (Participants) | 0 | 171 | 193
  Anti-varicella |  | 168 | 187

4. Primary Outcome: Number of Subjects With Vaccine Response for Anti-rubella Antibodies in HAV+MMR+V and MMR+V→HAV Groups
Description: Vaccine response is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination. Cut-off value assessed include 10 milli-international units per milliliter (mIU/mL).
Time Frame: 42 days following administration of M-M-R®II and VARIVAX®
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 247 | 271
Participants |  | 246 | 270

5. Secondary Outcome: Anti-measles, Anti-mumps, Anti-rubella and Anti-varicella Antibody Titers in HAV+MMR+V and MMR+V→HAV Groups
Description: Titers are given as geometric mean titers (GMTs).
Time Frame: 42 days following the administration of M-M-R®II and VARIVAX®
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 269 | 304
titers
  Anti-measles: number analyzed (Participants) | 0 | 269 | 301
  Anti-measles |  | 3218.3 [2940.9 to 3521.8] | 3136.3 [2922.0 to 3366.3]
  Anti-rubella |  | 88.3 [81.9 to 95.3] | 76.0 [70.7 to 81.7]
  Anti-varicella: number analyzed (Participants) | 0 | 218 | 260
  Anti-varicella |  | 281.7 [246.7 to 321.8] | 286.9 [252.1 to 326.5]
  Anti-mumps: number analyzed (Participants) | 0 | 244 | 276
  Anti-mumps |  | 215.7 [190.9 to 243.7] | 170.3 [152.2 to 190.5]

6. Secondary Outcome: Anti-hepatitis A Virus (HAV) Antibody Concentrations in HAV and HAV+MMR+V Groups
Description: Concentrations are given as geometric mean concentrations (GMCs).
Time Frame: 42 days following the first dose of Havrix®
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 228 | 0 | 306
milli-international units per milliliter | 43.1 [37.9 to 49.1] |  | 43.5 [39.3 to 48.2]

7. Secondary Outcome: Number of Subjects With Anti-hepatitis A Virus (HAV) Antibody Concentration Equal or Above the Cut-off Value in HAV and HAV+MMR+V Groups
Description: Anti-HAV antibody cut-off value assessed include 15 milli-international units per millilitre (mIU/mL).
Time Frame: 42 days following the first dose of Havrix®
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 228 | 0 | 306
Participants | 194 |  | 276

8. Secondary Outcome: Anti-hepatitis A Virus (HAV) Antibody Concentrations in MMR+V→HAV Group
Description: Concentrations are given as geometric mean concentrations (GMCs).
Time Frame: 31 days following the second dose of Havrix®
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results from MMR+V→HAV Group.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 237 | 0
milli-international units per milliliter |  | 1770.3 [1569.9 to 1996.4] |

9. Secondary Outcome: Number of Subjects With Anti-hepatitis A Virus (HAV) Antibody Concentrations Above the Cut-off Value in MMR+V→HAV Group
Description: Anti-HAV antibody cut-off value assessed include 15 milli-international units per millilitre (mIU/mL).
Time Frame: 31 days following the second dose of Havrix®
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 237 | 0
Participants |  | 237 |

10. Secondary Outcome: Number of Subjects With Vaccine Response to Havrix®
Description: Vaccine response was defined as: 1) a detectable anti-hepatitis A virus (HAV) antibody concentration 31 days following the second dose in subjects who were initially seronegative; and 2) a 2-fold increase in anti-HAV antibody concentrations above the pre-study concentration 31 days following the second dose in subjects who were initially seropositive.
Time Frame: 31 days following the second dose of Havrix®
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 194 | 224 | 259
Participants | 192 | 224 | 257

11. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, rash (local), redness and swelling.
Time Frame: During the 4-day period following each dose of vaccine
Population: Analysis was performed on the Total Vaccinated cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 304 | 411 | 419
Participants
  Pain | 103 | 162 | 187
  Rash (local) | 0 | 3 | 4
  Redness | 97 | 149 | 151
  Swelling | 45 | 70 | 82

12. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever, irritability, loss of appetite and rash (general).
Time Frame: During the 4-day period following each dose of vaccine
Population: Analysis was performed on the Total Vaccinated cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 304 | 424 | 411
Participants
  Drowsiness | 95 | 179 | 178
  Fever | 54 | 110 | 80
  Irritability | 144 | 238 | 216
  Loss of appetite | 94 | 170 | 154
  Rash (general) | 5 | 7 | 10

13. Secondary Outcome: Number of Subjects Reporting Measles, Mumps, Rubella and Varicella Specific Solicited General Adverse Events
Description: Specific adverse events assessed include papules, vesicles, crusts, parotid/salivary gland swelling and suspected signs of meningitis/febrile seizures.
Time Frame: During the 43-day period following each dose of vaccine
Population: Analysis was performed on the Total Vaccinated cohort, on subjects from MMR+V→HAV and HAV+MMR+V groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 0 | 455 | 462
Participants
  Papules |  | 23 | 23
  Vesicles |  | 17 | 17
  Crusts |  | 12 | 12
  Parotid/salivary gland swelling |  | 0 | 1
  Suspected signs of meningitidis/febrile seizures |  | 1 | 2

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms
Time Frame: During the 31-day period following each dose of vaccine
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 324 | 455 | 462
Participants | 186 | 286 | 249

15. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the Active Phase (from Day 0 up to Day 31 after the second dose) and the Extended Safety Follow-up Phase of the study (from Day 31 after the second dose up to study end)
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 324 | 455 | 462
Participants
  Active Phase | 1 | 6 | 5
  Extended Safety Follow-up Phase: number analyzed (Participants) | 287 | 376 | 395
  Extended Safety Follow-up Phase | 6 | 6 | 11

16. Secondary Outcome: Number of Subjects Reporting New Chronic Illnesses
Description: New Chronic illnesses include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: as for outcome 15
Population: Analysis was performed on the Total Vaccinated cohort (for the Active Phase) and the Extended Safety Follow-up cohort (for the Extended Safety Follow-up Phase).
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 324 | 455 | 462
Participants
  Active Phase | 0 | 0 | 0
  Extended Safety Follow-Up Phase: number analyzed (Participants) | 287 | 376 | 395
  Extended Safety Follow-Up Phase | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects Reporting Medically Significant Events
Description: Medically significant events include, but are not limited to, diabetes, autoimmune disease, asthma, allergies and/or conditions prompting emergency room or physician office visits that are not related to well-child care, vaccination or common acute illnesses (e.g., upper respiratory infection, otitis media, pharyngitis, gastroenteritis, injury and visits for routine physical examination).
Time Frame: as for outcome 15
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Number analyzed (Participants) | 324 | 455 | 462
Participants
  Active Phase | 0 | 0 | 0
  Extended Safety Follow-Up Phase: number analyzed (Participants) | 287 | 376 | 395
  Extended Safety Follow-Up Phase | 0 | 0 | 0

ADVERSE EVENTS:
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available.
  Events collected by non-systematic method are reported for the Total Vaccinated Cohort
Arm/Group | HAV Group | MMR+V→HAV Group | HAV+MMR+V Group
Serious Adverse Events (participants affected / at risk) | 7/324 | 12/455 | 16/462
Other Adverse Events (participants affected / at risk) | 251/324 | 366/455 | 363/462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HAV Group (N=324) | MMR+V→HAV Group (N=455) | HAV+MMR+V Group (N=462)
Dehydratation (Metabolism and nutrition disorders) | 2 | 1 | 2
Bronchiolitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mental retardation (Nervous system disorders) | 0 | 0 | 1
Autism (Nervous system disorders) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Breathing-related sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HAV Group (N=324) | MMR+V→HAV Group (N=455) | HAV+MMR+V Group (N=462)
Otitis media (Infections and infestations) | 35 | 79 | 65
Pyrexia (General disorders) | 34 | 68 | 56
Upper respiratory tract infection (Infections and infestations) | 31 | 64 | 58
Diarrhoea (Gastrointestinal disorders) | 16 | 39 | 22
Teething (Gastrointestinal disorders) | 25 | 24 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 20 | 23
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 20 | 22 | 17
Nasopharyngitis (Infections and infestations) | 19 | 19 | 19
Vomiting (Gastrointestinal disorders) | 14 | 30 | 12
Papules (General disorders) | 0/0 | 23 | 23
Drowsiness (General disorders) | 95/304 | 179/411 | 178/424
Fever (General disorders) | 54/304 | 110/411 | 80/424
Irritability (General disorders) | 144/304 | 238/411 | 216/424
Loss of appetite (General disorders) | 94/304 | 170/411 | 154/424
Pain (General disorders) | 103/304 | 162/411 | 187/419
Redness (General disorders) | 97/304 | 149/411 | 151/419
Swelling (General disorders) | 45/304 | 70/411 | 82/419

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.